CLINICAL TRIAL: NCT06632340
Title: Effect of Tumor Base Size on Recurrence and Progression in Non-muscle Invasise Bladder Cancer
Brief Title: Effect of Tumor Base Size in Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Bedirhan Bayraktar, medical doctor, Ankara Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCTB2024
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): tumor base size <2 cm
  Interventions: Procedure: TUR-BT
- Group 2 (Other): tumor base size >2 cm
  Interventions: Procedure: TUR-BT

INTERVENTIONS:
Procedure: TUR-BT — Transurethral resection of bladder tumor

SUMMARY:
Investigators aim to investigate the effect of the size of the base of the tumor in contact with the bladder mucosa on recurrence and progression in non-muscle invasive bladder tumors.

DETAILED DESCRIPTION:
Between March 2021 and September 2023, 130 patients who applied to our clinic with complaints of hematuria, dysuria, and suprapubic pain, and who were diagnosed with bladder tumor by imaging methods and underwent TUR-MT were included in the study. The groups were compared in terms of age, gender, smoking, ASA, comorbidities, BMI and the number of tumors, size, stage as intraoperative and postoperative data. Patients with tumor base size <2 cm were classified as Group

1, while with tumor base size ≥2 cm were classified as Group 2. Kaplan Meier survival analysis without recurrence and without progression were performed after comparing the groups in terms of recurrence and progression.

ELIGIBILITY:
Inclusion Criteria:

* Bladder Tumor

Exclusion Criteria:

* Invasive Bladder Tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | 2 year

SECONDARY OUTCOMES:
progression | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)